CLINICAL TRIAL: NCT06040008
Title: Investigating the Impact of Environmental Factors on the Transcriptomics Profile in Healthy Individuals: Comparison of PaxGene RNA Tube and Dried-Blood-Spot Filter Card (CENTOCARD®)
Brief Title: Investigating the Impact of Environmental Factors on the Transcriptomics Profile in Healthy Individuals
Acronym: IMEN
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: IS 01-2023
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- healthy volunteers: Healthy status is defined by the absence of evidence of any active or chronic disease at the beginning of the study
  Interventions: Genetic: blood collection

INTERVENTIONS:
Genetic: blood collection — * 3 blood collections over a period of 6 weeks
  * V0 - Inclusion
  * V1 - 3 weeks ± 14 days
  * V2 - 3 weeks ± 14 days
  * 1 EDTA 4 ml tube, 1 PAXgene RNA tube 2,5 ml and drops of blood from finger-prick are taken at each visit
  * Clinical information obtained at each visit

SUMMARY:
Changes in biology will be reflected by changes in the composition of Ribonucleic acid (RNA) in the blood. An example of that would be environmental changes, e.g. diet, acute illness, temperature. The main goal of this study is to study the impact of environmental changes in blood transcriptomics in healthy individuals over time.

DETAILED DESCRIPTION:
The project is aiming to evaluate the impact of environmental changes on the blood transcriptome and to assess the feasibility of different sample collection materials for this purpose. Transcriptome from EDTA-DBS. Performing RNAseq from EDTA-DBS, Finger-Prick- DBS and PAXgene RNA tubes has resulted in different levels of analytical "background noise".

To measure the reflection of this noise, we aim to collect and evaluate blood samples of participating healthy individuals on different time points, to discover how suitable, the DBS is in detecting changes caused by environmental factors (diet, acute disease, temperature). The environmental factors should have variable severity of changes.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, informed consent is obtained from the subject before enrollment in the study
* The subject is 18 years or older (≥18 years)
* Healthy participants, as declared by the subject
* Healthy status is defined by the absence of evidence of any active or chronic disease at the beginning of the study
* Available to participate for the planned duration of the study for which the screening is being done

Exclusion Criteria:

* • The subject had any clinically significant disease

  * Any clinically relevant history or the presence of e.g., respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, etc. chronic disease
  * Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
  * A condition in which repeated blood draws poses more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access
  * In the opinion of the investigator, subject is at high risk of non-compliance and is unsuitable in any other way to participate in this study
  * No informed consent obtained from the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy participants
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
study the impact of environmental changes in blood transcriptomics | 12 months
  Changes in biology will be reflected by changes in the composition of Ribonucleic acid (RNA) in the blood. An example of that would be environmental changes, e.g. diet, acute illness, temperature.

SECONDARY OUTCOMES:
different sample collection materials | 12 months
  The secondary goal is to evaluate the feasibility of different sample collection materials. RNA collected from PAXgene RNA tubes is a gold standard for RNA extraction from blood.
  However, CENTOGENE devised an alternative method to obtain RNA from CentoCard® (or Dried-Blood-Spot card/DBS). There is a systematic difference between these methods regarding the extraction and depletion of hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Böttcher, MD, Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- Centogene GmbH, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No